CLINICAL TRIAL: NCT04736225
Title: Effects of the Insulin Self-titration Education on Glycemic Control in Type 2 Diabetes Mellitus Patients: A Quasi-Experimental Study
Brief Title: Effects of the Insulin Self Titration Education for Type 2 Diabetes Mellitus Patients
Acronym: ISTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Chiayi Christian Hospital (Other)
Responsible Party: Principal Investigator, Tsae Jyy, Wang, Principal Investigator, National Taipei University of Nursing and Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CCYCH-099034
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Type2 Diabetes
Keywords: Blood Glucose Self-Monitoring; Type 2 Diabetes Mellitus; Self Efficacy; Self Care,
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ISTE Group (Experimental): This program includes a 60-min small-group lesson, a 20-min individual instruction. The education program's goal is to teach patients to self-titrate their insulin doses every six days to maintain their six-day average blood glucose levels < 120 mg/dl
  Interventions: Other: Insulin Self-Titration Education Program
- Non-ISTE Group (Placebo Comparator): The usual care (a 15-min individual education) was giving at the Diabetes Health Education Center. They were taught how to self-inject insulin and test and record their before-breakfast and before-dinner blood glucose levels daily at home.
  Interventions: Other: Insulin Self-Titration Education Program

INTERVENTIONS:
Other: Insulin Self-Titration Education Program — The program contents of instruction included blood glucose self-monitoring, types of insulin, insulin self-administration, insulin dose titration, hyperglycemia or hypoglycemia self-management, diet, and exercise.a 20-min one-on-one training session from a nurse on how to self-titrate the insulin dose. The participants were taught to monitor their before-breakfast and before-dinner blood glucose levels at home and adjust their insulin doses accordingly.

SUMMARY:
The purpose of the study was to evaluate the effects of an insulin self-titration education program on glycemic control, self-efficacy, and self-care behaviors in patients with type 2 diabetes. The quasi-experimental design was adapted. A convenient sample of 120 patients with insulin-treated type 2 diabetes was recruited from a general hospital in Taiwan. Among them, 60 were in the insulin self-titration group, and 60 were in the comparison group. Data on glycated hemoglobin (HbA1C), self-efficacy, and self-care behavior were collected at baseline, three-month, and six-month follow-up. The study instruments included the Insulin Diabetes Management Self-Efficacy Questionnaire and Diabetes Self-Care questionnaire.

DETAILED DESCRIPTION:
Sixty patients with insulin-treated type 2 diabetes were recruited as the intervention participants and enrolled in the insulin self-titration program. Sixty propensity score-matched patients treated with traditional insulin therapy without self-titration were recruited as the control participants. Data on HbA1C and hypoglycemia were collected at baseline and during follow-ups at three and six months. Data on self-efficacy and self-care were collected at the six-month follow-up using self-report questionnaires.

The inclusion criteria were recruited: (1) age ≥ 18 years; (2) diagnosis of type 2 diabetes; (3) treatment with insulin injection for > six months; (4) HbA1C > 7.5% in the last three months; and (5) ability to communicate in Mandarin or Taiwanese.

The insulin self-titration education program includes a 60-min small-group lesson, a 20-min individual instruction. Patients in the comparison group received usual care at the Diabetes Health Education Center. During a 15-min individual education, these patients were taught how to self-inject insulin and test and record their before-breakfast and before-dinner blood glucose levels daily at home Data on glycated hemoglobin (HbA1C) and the number of hypoglycemia were collected at baseline, three-month, and six-month follow-up. Data on self-efficacy and self-care were collected at the six-month follow-up, using the self-reported questionnaires. The study was approved by the institutional review board of the hospital where the data were collected.

Data were analyzed by using the SPSS 21.0 software. Descriptive analyses were used to describe the research variables. Chi-Square and independent t-test were used to analyze the baseline equilibriums between the two groups. Independent t-tests were used to analyze between-group differences in HbA1C at each time point. A generalized estimating equation (GEE) was used to analyze between-group differences in HbA1C change over time. The independent t-test was used to analyze the difference between the two groups of participants in the post-testing diabetes self-efficacy and self-care.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* diagnosis of type 2 diabetes
* treatment with insulin injection for > six months
* HbA1C > 7.5% in the last three months
* ability to communicate in Mandarin or Taiwanese

Exclusion Criteria:

* non

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2011-07-30 (Actual); Study Completion 2011-07-30 (Actual)

PRIMARY OUTCOMES:
HbA1C | six-month follow-up
  HbA1c was measured by a 3cc venous blood sample was and analyzed with the Tosoh G8 HPLC Analyzer.

SECONDARY OUTCOMES:
self-efficacy | six-month follow-up
  The Chinese version of the Insulin Management Diabetes Self-Efficacy Scale (IMDSES) was used to assess a participant's degree of confidence in the ability of self-controlled diabetes. The 28-item scale includes six subscales: general self-efficacy, dietary self-efficacy, insulin self-efficacy, blood glucose monitoring self-efficacy, exercise self-efficacy, and foot self-efficacy. Each item is rated on a scale from 0 (completely unsure) to 100 (very sure). The average score of all items represents the scale sore, with a possible range of 0 to 100. The higher the score the better the self-efficacy. In this study, the Cronbach's α of this scale was 0.89, and the Cronbach's α value of each sub-scale was between 0.69 and 0.95.
self-care behavior | six-month follow-up
  The Chinese version of the revised Diabetes Self-Care Scale (DSC) was used to measure a participant's self-care behavior. The 28-item scale includes six subscales: general self-care, self-care for diet, self-care for insulin adjustment, self-care for blood glucose monitoring, self-care for exercise, and self-care for the feet. Each item is rated on a scale from 0 (not done at all) to 100 (completely done). The average score of all items represents the scale score, with a possible range of 0 to 100. The higher the score the better the self-care behavior. In this study, the Cronbach's α of this scale was 0.89, and the Cronbach's α value of each subscale was between 0.69 and 0.86.

CONTACTS AND LOCATIONS:
Overall Officials: Tsae-Jyy Wang, Principal Investigator — National Taipei University of Nursing and Health Science

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davies MJ, D'Alessio DA, Fradkin J, Kernan WN, Mathieu C, Mingrone G, Rossing P, Tsapas A, Wexler DJ, Buse JB. Management of Hyperglycemia in Type 2 Diabetes, 2018. A Consensus Report by the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetes Care. 2018 Dec;41(12):2669-2701. doi: 10.2337/dci18-0033. Epub 2018 Oct 4. PMID 30291106
- [Result] Tomah S, Mahmoud N, Mottalib A, Pober DM, Tasabehji MW, Ashrafzadeh S, Hamdy O. Frequency of self-monitoring of blood glucose in relation to weight loss and A1C during intensive multidisciplinary weight management in patients with type 2 diabetes and obesity. BMJ Open Diabetes Res Care. 2019 Jul 29;7(1):e000659. doi: 10.1136/bmjdrc-2019-000659. eCollection 2019. PMID 31413841
- [Result] Misra A, Patel M, Agarwal P, Lodha S, Tandon N, Magdum M, Yajnik C, Ghosh R, Walekar A. Effectiveness and Safety of Physician-Led Versus Patient-Led Titration of Insulin Glargine in Indian Patients with Type 2 Diabetes Mellitus: A Subanalysis of the Asian Treat to Target Lantus Study (ATLAS). Diabetes Technol Ther. 2019 Nov;21(11):656-664. doi: 10.1089/dia.2019.0037. Epub 2019 Aug 9. PMID 31335198